CLINICAL TRIAL: NCT03715712
Title: Comparison of Individualized vs Standard Blood Pressure Target on the Postoperative Myocardial Injury in High Risk Patients Undergoing Non-cardiac Surgery- a Randomized Non-inferiority Trial
Brief Title: NORepinephrine-Maintaining-individuaALIZEd Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NORMALIZE
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Perioperative Myocardial Injury; Blood Pressure; Non-cardiac Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Experimental): Standardized blood pressure management with a target of mean blood pressure greater than 65mmHg and systolic blood pressure lower than 160mmHg
  Interventions: Other: standardized blood pressure management
- Individualized (Active Comparator): Individualized blood pressure management of 20% within the preoperative ward blood pressure
  Interventions: Other: Individualized blood pressure management

INTERVENTIONS:
Other: standardized blood pressure management — Standardized blood pressure management of a mean blood pressure > 65mmHg and a systolic blood pressure of < 160mmHg using norepinephrine continuous infusion
  Arms: Standard
Other: Individualized blood pressure management — Individualized blood pressure management of 20% within the preoperative ward blood pressure using norepinephrine continuous infusion
  Arms: Individualized

SUMMARY:
This study compares the effect of individualized vs standard blood pressure management on postoperative myocardial injury in high-risk patients undergoing non-cardiac surgery by measuring the hs-cTnT levels. Continuous norepinephrine infusion is used to target a mean pressure of greater than 65mmHg and a systolic pressure less than 160mmHg in the standardized group while the target is 20% within the ward blood pressure in the individualized group. The pre- and postoperative hs-cTnT levels to detect myocardial injury are compared between the two groups.

DETAILED DESCRIPTION:
Managing the blood pressure preoperatively is important in high-risk patients because hypotension can lead to perioperative myocardial injury. It has been reported that a systolic pressure of less than 50-55mmHg or greater than 40% decrease can lead to cardiac complications. The mechanism of hypotension leading to postoperative myocardial injury is due to hypoperfusion and ischemic reperfusion injury.

In this randomized controlled study, the blood pressure for participants in the standardized group is maintained as follows: mean blood pressure greater than 65mmHg and systolic blood pressure less than 160mmHg. The individualized group participants' blood pressure is maintained at a target of 20% within the preoperative ward blood pressure. Anesthesia and intraoperative management are the same in both groups to target a bispectral index level of 50. In order to quantitatively measure the myocardial injury, high sensitive cardiac troponin T (hs-cTnT) will be measured pre- and postoperatively. A level greater than 14ng/dl has been reported to be associated with myocardial injury and mortality. The objective of this study is to show that the standardized protocol of maintaining a mean pressure greater than 65mmHg is non inferior to the individualized management in terms of postoperative myocardial injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general or urologic surgeries under general anesthesia at Seoul National University Hospital
* high-risk patients with a revised cardiac risk index of at least 2 points or more

Exclusion Criteria:

* severely uncontrolled hypertension (systolic blood pressure ≥ 180mmHg or mean blood pressure ≥ 110)
* severely uncontrolled hypotension (systolic blood pressure < 80mmHg)
* arrhythmias with symptoms or use of pacemaker
* transplantation surgery
* acute or decompensated heart failure
* acute coronary syndrome
* sepsis
* end stage renal disease (GFR <30ml/min/1.73m2)
* contraindications of norepinephrine infusion

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of postoperative myocardial injury | baseline and postoperative day 1
  the change of hs-cTnT levels

SECONDARY OUTCOMES:
hospital LOS | 1 month
  hospital length of stay
ICU LOS | 1 month
  ICU length of stay
in hospital mortality | 1 month
  in hospital mortality
Amount of norepinephrine used | intraoperative
  total amount of norepinephrine used
intraoperative vital signs | intraoperative
  blood pressure, heart rate, ECG, stroke volume, stroke volume variation, bispectral index
acute myocardial complications | 1 month
  chest pain, dyspnea, edema, acute coronary syndrome
acute kidney injury | postoperative 48 hours
  serum creatinine increase and urine output

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea